CLINICAL TRIAL: NCT02770040
Title: PREDICT UC: Optimising Infliximab Induction Therapy for Acute Severe Ulcerative Colitis
Brief Title: Optimising Infliximab Induction Therapy for Acute Severe Ulcerative Colitis
Acronym: PREDICT UC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Austin Health (Other Government)
Collaborators: University of Melbourne (Other)
Responsible Party: Principal Investigator, Dr Peter De Cruz, Head of Inflammatory Bowel Disease Unit, Austin Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREC/14/Austin/595
Record Dates: First submitted 2016-05-09; First posted 2016-05-12 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Ulcerative Colitis
Keywords: Acute Severe Ulcerative Colitis; Steroid Refractory Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intensified Infliximab Induction (Active Comparator): Infliximab 10mg/kg at Week 0 and Week 1
  Interventions: Drug: Infliximab
- Accelerated Infliximab Induction (Active Comparator): Infliximab 5mg/kg at Week 0, Week 1 and Week 3
  Interventions: Drug: Infliximab
- Standard Infliximab Induction (Active Comparator): Infliximab 5mg/kg at Week 0, Week 2 and Week 6
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — INFLIXIMAB (REMICADE) in the form of a freeze-dried compound is conditioned in 100mg vials. Treatment will first be reconstituted in 250ml isotonic saline solution and infused
  Other Names: Remicade

SUMMARY:
The purpose of this study is to identify whether an Accelerated or Intensified Infliximab induction regimen is superior to Standard induction in Acute Severe Ulcerative Colitis in an open label multi-centre randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Diagnosis of Ulcerative Colitis
* Acute Severe Colitis according to the Truelove and Witt's Criteria
* Steroid refractory according to the Oxford Criteria

Exclusion Criteria:

* Participant unable to consent for themselves
* Indication for immediate surgery (acute abdomen, perforation of the bowel, haemorrhage)
* Crohn's disease
* Participants with enteric infection confirmed on stool microscopy, culture or toxin
* Haemodynamic instability (mean arterial pressure <60) and not responsive to fluids
* Participants with clinically significant Cytomegalovirus infection (positive inclusion bodies, immunohistochemistry and signs of viraemia such as fever and abnormal liver function tests)
* Participants who are pregnant or currently breast-feeding
* Participants with current malignancy, excluding basal cell carcinoma
* Participants with flat low or high grade colonic dysplasia; sporadic adenomas permitted
* Participants with serious co-morbidities including: Immunodeficiency; Myocardial infarction or acute stroke within the last 3 months; Moderate or severe heart failure (New York Heart Association class III or IV); Active or suspected tuberculosis; Renal failure; Hepatic failure; other severe infections
* Participants with history of hypersensitivity to infliximab or infliximab biosimilar
* Participants who have received other immunosuppressive agents including but not limited to: Anti-TNF therapies within 3 months of screening (Infliximab, Infliximab biosimilar, Golimumab, Etanercept, Certolizumab or Adalimumab); Anti-integrins (Vedolizumb, Etrolizumab) within 4 months of screening; Calcineurin inhibitors (Cyclosporine, Tacrolimus) within 4 weeks of screening; T or B cell depleters (Rituximab, Alemtuzumab) within 12 months of screening; other investigational agents (eg. Ustekinumab) within 6 months of screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Clinical response by day 7 | Day 7
  Defined as a reduction in the Lichtiger score below 10 with a decrease of at least 3 points and an improvement in rectal bleeding and stool frequency to ≤4 per day

SECONDARY OUTCOMES:
Time to clinical response | Up to 3 months
Colectomy by Day 7 | From Day 0 to Day 7

OTHER OUTCOMES:
Colectomy free survival at 1 month, 3 months and 12 months | Up to 12 months
  Effect estimates between different dose regimens
Steroid free remission at 3 months | Day 90
  Defined as a Mayo disease activity index score ≤2 with an endoscopic subscore ≤1
Endoscopic remission rates at 3 and 12 months | Up to 12 months
  Defined by a Mayo endoscopic subscore of ≤1

CONTACTS AND LOCATIONS:
Overall Officials: Peter De Cruz, MBBS PhD FRACP, Principal Investigator — Austin Health, Melbourne; Matthew C Choy, MBBS BMedSci FRACP, Principal Investigator — Austin Health, Melbourne
Locations (1):
- Austin Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choy MC, Li Wai Suen CFD, Con D, Boyd K, Pena R, Burrell K, Rosella O, Proud D, Brouwer R, Gorelik A, Liew D, Connell WR, Wright EK, Taylor KM, Pudipeddi A, Sawers M, Christensen B, Ng W, Begun J, Radford-Smith G, Garg M, Martin N, van Langenberg DR, Ding NS, Beswick L, Leong RW, Sparrow MP, De Cruz P. Intensified versus standard dose infliximab induction therapy for steroid-refractory acute severe ulcerative colitis (PREDICT-UC): an open-label, multicentre, randomised controlled trial. Lancet Gastroenterol Hepatol. 2024 Nov;9(11):981-996. doi: 10.1016/S2468-1253(24)00200-0. Epub 2024 Sep 2. PMID 39236736